CLINICAL TRIAL: NCT03556176
Title: The Influence of 5-HTTLPR and BDNF Polymorphisms on Anxiety and Mood After Acute Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Luiz Carlos Bandeira Santos Júnior, Professor, Universidade Federal de Goias
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2.331.601
Record Dates: First submitted 2018-05-08; First posted 2018-06-14 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Polymorphisms; Exercise; Mood
Keywords: Anxiety; Mood; Physical activity; Polymorphisms
MeSH Terms: conditions — Motor Activity; Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-HTTLPR or BDNF polymorphisms (Active Comparator)
  Interventions: Behavioral: Exercise; Behavioral: Quiet rest
- Control ( without 5-HTTLPR or BDNF polymorphisms ) (Active Comparator)
  Interventions: Behavioral: Exercise; Behavioral: Quiet rest

INTERVENTIONS:
Behavioral: Exercise — Three exercises sessions - 30 min (light: 45 - 50%, moderate: 65 -70% and vigorous: 85 - 90% Heart Rate Maximal).
Behavioral: Quiet rest — Quiet rest during 30 min

SUMMARY:
The Influence of 5-HTTLPR and BDNF Polymorphisms on Anxiety and Mood After Acute Exercise.

Introduction: The 5-HTTLPR (SLC6A4) and BDNF (Val66Met) polymorphism presents an action on the modulation of human behavior and has received great attention as a risk factor for several psychiatric disorders. In recent years, a growing number of studies have evaluated the association between these polymorphisms and personality traits related to anxiety and depression. Objectives: To determine the frequencies of 5-HTTLPR and BDNF polymorphisms in a college students population; To determine the influence of 5-HTTLPR and BDNF polymorphisms on mood states and anxiety after acute physical exercise. Material and Methods: Four hundred (400) College students will be assessed.

In the first phase of the study, the following procedures will be performed: Screening, Aerobic Fitness Assessment (Step Test), Questionnaires (PAR-Q, Habitual Physical Activity Level, Beck Anxiety and Depression Scale, State-Trait Anxiety, and Perceived Stress Scale), blood sample collection and genotyping. In the second phase of the study, two (2) groups with or without polymorphisms will be selected (for each gene). These groups will be submitted to four conditions (three experimental conditions and one control condition), carried out randomly and separated by an interval of 1 week. In the experimental Conditions the volunteers will perform treadmill exercises sessions (30 minutes) in three different intensities (light, moderate and vigorous) and will respond to the Borg Scale at 10, 20 e 30 minutes. In the control condition the volunteers will be instructed to remain seated (quiet rest), relaxed and silent for 30 minutes. In both conditions, the volunteers will complete the Profile of Mood States (POMS) and State-Anxiety (STAY), 05 (five) minutes before and, 5 (five) and 20 (twenty) minutes following the interventions.

ELIGIBILITY:
Inclusion criteria:

* 18-30 years of age;
* able to perform physical activities;

Non-inclusion criteria:

* history of cardiovascular or respiratory diseases;
* smoking;
* use of psychiatric drugs;
* psychotherapy treatment in the last six months.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Response of mood states after interventions | Change from 5 minutes before the treatments to 5 and 20 minutes after three exercise intensities and quiet rest
  The POMS questionnaire is an instrument to evaluate mood states. It has 65 items and 6 domains: tension-anxiety, depression, anger-hostility, vigour-activity, fatigue, and confusion- bewilderment. The total mood disturbance score is derived by subtracting the vigour-activity score from the the sum of scores from the other subscales. The iceberg profile is characterized by low raw scores on the tension, depression, anger, fatigue, and confusion scales and above norms (the "water line") on vigor.
Response of anxiety after interventions | Change from 5 minutes before the treatments to 5 and 20 minutes after three exercise intensities and quiet rest
  Anxiety Inventory-STAI trait-state. The scales encompasses 20 items and provides a one-dimensional measurement of anxiety. Range of scores for each subtest is 20-80, the higher score indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms.

SECONDARY OUTCOMES:
Evaluation safety or possible risk of exercising | baseline
  The Physical Activity Readiness Questionnaire (PAR-Q) was originally designed as a screening questionnaire to be self-administered before beginning physical activity. It has been designed to identify the small number of adults for whom physical activity may be inappropriate or those who should have medical advice concerning the type of activity most suitable for them.The people who to answer yes to one or more of seven questions will be advised to consult their doctors before increasing their physical activity. Those who to answer no to all questions will be included in the protocol study.
Habitual Physical Activity Level | Baseline
  Habitual Physical Activity Level (BAECKE):The Baecke Questionnaire was developed to measure habitual physical activity. The questionnaire includes items about household activities, sport, and leisure time activities over the past year. The Sport Index is divided into four categories (<1 h; 1-2 hrs; 2-3 hrs; 3-4 hrs and > 4 hrs) and each of these categories has an appropriate coefficient (0.5; 1.5; 2.5; 3.5 and 4.5) Usual daily activity and leisure activity are scored in a range of from 0 to 5. Global PA will be the sum of 3 indexes.
Evaluation of depression and anxiety symptoms | Baseline
  Beck Inventory Anxiety and Depression: The Beck Depression and Anxiety Inventory consists of a self-report questionnaires. These instruments are used to measure the severity of depressive and anxiety episodes.These instruments are widely used by health professionals and researchers in a variety of clinical and research settings.
  In the Beck Depression Inventory normal score are between 0 and 15; medium depression scores from 15 to 20 (dysphoria), and high depression scores over 20, and in the Beck Anxiety Inventory: 0-9: normal to minimal anxiety;10-18: mild to moderate anxiety;19-29: moderate to severe anxiety and 30-63: severe anxiety.
Estimation the aerobic capacity | Baseline
  McArdle Step Test was developed to estimate the aerobic capacity of university students. For the test the individual must ascend and descend a step during 3 min with different stepping rates for women and men (22 and 24 steps/min, respective
Detection of the polymorphism in the SLC6A4 | Baseline
  The detection of the polymorphism in the SLC6A4 gene will be done by the PCR-RFLP method: restriction fragment length polymorphism (RFLP), in which the PCR amplification of the flanking region of the SNP is followed by the digestion reaction with a specific restriction enzyme.
  The polymorphism of the SLC6A4 gene will be determined by the Polymerase Chain Reaction (PCR) and subsequent gel electrophoresis. PCR will be performed with the following primers forward (GGCGTTGCCGCTCTGAATGC) and reverse (GAGGGACTGAGCTGGACAACCAC).
Detection of the polymorphism BDNF Val66Met SNP rs6265 genotype (G196A) | Baseline
  The BDNF Val66Met SNP rs6265 genotype (G196A) will be obtained, using a polymerase chain reaction-restriction fragment length polymorphism (PCR-RFLP) method with forward (5'-ACTCTGGAGAGCGTGAAT-3') and reverse (5'-ATACTGTCACAC ACGCTC-3') primers, and further digestion of the PCR product with NlaIII enzyme (Cat. No. R0125S, New England Biolabs).
  From the five possible restriction fragments for this Val66Met amplicon, the genotype will be identified by the size and distribution of three bands: 243 bp for the G variant (Val), 168 bp and 75 bp bands for the A variant (Met), and these three bands for GA heterozygotes (Val/Met), on 2.5% (w/v) agarose gel electrophoresis.

CONTACTS AND LOCATIONS:
Locations (1):
- UFG, Jatai, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Undecided